CLINICAL TRIAL: NCT04968951
Title: REFOCUS: Refined Fecal Microbiota Transplantation (FMT) Delivered by Oral Capsules for Induction of Remission in Mild to Moderate Ulcerative Colitis - a Phase I Study
Brief Title: Refined Fecal Microbiota Transplantation (FMT) for Ulcerative Colitis (UC)
Acronym: REFOCUS
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: insufficient funding
Sponsor: Ari M Grinspan (Other)
Responsible Party: Sponsor-Investigator, Ari M Grinspan, Associate Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 18-1464
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis; FMT; Fecal Microbiota Transplant
Keywords: FMT; Fecal Microbiota Transplantation; Fecal Microbiota Transplant; Fecal Matter Transplant; Ulcerative colitis; UC
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Metronidazole; Vancomycin; Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups. One group will be assigned to receive pre-treatment with antibiotics before Fecal Microbiota Transportation. The other group will be assigned to receive pre-treatment without antibiotics (with placebo) before Fecal Microbiota Transplantation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Antibiotics and placebo will be disguised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMT with Antibiotics (Active Comparator): Participants will receive antibiotics before receiving Fecal Microbiota Transplantation
  Interventions: Drug: Metronidazole; Drug: Vancomycin; Biological: Fecal Microbiota Transplantation
- FMT with placebo (Placebo Comparator): Participants will receive placebo before receiving Fecal Microbiota Transplantation
  Interventions: Drug: Placebo; Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Metronidazole — Antibiotic treatment - 250 mg every 6 hrs for 5 days
  Other Names: Flagyl
  Arms: FMT with Antibiotics
Drug: Placebo — Placebo treatment
  Arms: FMT with placebo
Drug: Vancomycin — Antibiotic treatment - 125 mg every 6 hrs for 5 days
  Arms: FMT with Antibiotics
Biological: Fecal Microbiota Transplantation — Encapsulated biologically active human fecal material (donor stool) is provided in capsule form. The fecal material is homogenized with sterile saline, then pelleted and re-suspended in sterile saline/40% glycerol. Participants will receive 15 FMT capsules per day for 3 consecutive days. Capsule are to be swallowed under direct supervision.
  Other Names: FMT

SUMMARY:
The researchers intend to prospectively study the safety, clinical efficacy and microbial outcomes in patients with recently diagnosed UC with FMT capsule therapy derived from pre-defined donors. Donors will be specifically screened for Fusobacterium and Sutterella species as well as for global diversity. It is unknown if treatment with antibiotics before FMT improves the engraftment and/or efficacy of FMT in UC, therefore the researchers plan to randomize subjects to receive pre-treatment with antibiotics or not before FMT therapy. The research team enroll patients from The Susan and Leonard Feinstein IBD Center and our established early diagnosis clinic at Mount Sinai Hospital (MSH).

DETAILED DESCRIPTION:
This is an open-label two arm pilot study to measure the safety, microbiological and clinical impacts of FMT in patients with ulcerative colitis. The researchers will prospectively enroll 16 UC patients (up to 20 subjects accounting for subjects dropping out) with moderate-severe disease from one tertiary care referral center. The overall objective of the study is to collect robust clinical data and create a tissue repository including blood, stool and biopsies to understand the safety, efficacy and microbial changes FMT has on UC patients. The central hypothesis is that pre-defined oral capsule administered FMT is safe and effective for the treatment of UC.

Objectives: To determine the tolerability, feasibility, and safety of using fecal microbiota transplantation orally as an induction agent for patients with ulcerative colitis. To determine whether fecal microbiota transplantation (FMT) delivered via oral capsules can induce clinical remission in patients with mild to moderate ulcerative colitis. Assess whether pretreatment with antibiotics improves engraftment and efficacy of FMT in UC. To characterize the impact of orally administered FMT on the microbiota of patients with ulcerative colitis, particularly those changes associated with response or lack of response.

Study Outcomes: Clinical remission at Week 8, defined as: Steroid-free clinical remission (Total Mayo less 2) and Endoscopic remission (Mayo endoscopic subscore 0 or 1)

ELIGIBILITY:
* Adults aged 18 to 75 with UC, with initial diagnosis of UC >3 months prior to time of study enrollment visit
* Partial Mayo score of 4-10 with endoscopic subscore ≥2 on flexible sigmoidoscopy
* Permissible UC medications include oral or rectal administered mesalamines
* Corticosteroids must be discontinued at least 4 weeks before enrollment
* Documented negative C. difficile and GI PCR for enteric pathogens (BioFire) testing before commencement of fecal microbiota transplantation
* Previous documentation of ulcerative colitis based on colonoscopy/flexible sigmoidoscopy with compatible histology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an adverse | 8 Weeks
  Safety as measured by proportion of participants with an adverse event through week 8
Proportion of participants with a severe adverse | 8 Weeks
  Safety as measured by proportion of participants with a severe adverse event through week 8

SECONDARY OUTCOMES:
Number of patients requiring escalation of medical therapies | 8 weeks
  Number of patients requiring escalation of medical therapies based on clinical relapse. Clinical relapse is defined by requiring additional medical therapy.
Proportion of patients that achieve Mayo score 0 or 1 | 8 weeks
  Proportion of patients with initial Mayo 2/3 disease at flexible sigmoidoscopy that achieve endoscopic improvement (Mayo score 0 or 1). The Mayo Score is a composite of subscores (each rated 0-3) from four categories, including stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy or colonoscopy, and physician's global assessment, with a total score ranging from 0-12, with higher score indicating worse health outcomes.
Number of patients with endoscopic remission | 8 weeks
  Number of patients with endoscopic remission as defined by a Mayo score of 0
Change in Nancy score | 8 weeks
  Change in histological score assessed by the Nancy score. The Nancy score includes 3 histologic items that define 5 grades of activity: absence of significant histologic disease, chronic inflammatory infiltrate with no acute inflammatory infiltrate, mildly active disease, moderately active disease, and severely active disease. The Nancy index is defined by a 5-level classification ranging from grade 0 (absence of significant histological disease activity) to grade 4 (severely active disease). higher score indicating worse health outcomes.
Fecal calprotectin level | baseline and 8 weeks
  Mean change fecal calprotectin levels
C-reactive protein levels | baseline and 8 weeks
  Mean change C-reactive protein levels
Hemoglobin levels | baseline and 8 weeks
  Mean change hemoglobin levels
Albumin levels | baseline and 8 weeks
  Mean change albumin levels
ESR level | baseline and 8 weeks
  Mean change erythrocyte sedimentation rate (ESR)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Grinspan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available